CLINICAL TRIAL: NCT05305924
Title: Phase II Trial Of Fulvestrant Plus Abemaciclib In Er-Positive, Her2-Negative Metastatic Breast Cancer Immediately After Failure Of A Cdk4/6 Inhibitor
Brief Title: Fulvestrant+Abemaciclib With Run-In of Fulvestrant in Er-Positive, Her2-Negative Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Polly A. Niravath, MD, Professor of Medicine in Oncology, Academic Institute, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00028925
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: ER-Positive Breast Cancer; HER2-negative Breast Cancer
Keywords: Fulvestrant; Abemaciclib; CDK4/6 Inhibitor; Aromatase Inhibitor
MeSH Terms: interventions — abemaciclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fulvestrant plus Abemaciclib Arm with Fulvestrant Run-In (Experimental): A 1-month (28 days) run-in of fulvestrant will precede fulvestrant plus abemaciclib treatment. Fulvestrant at a dose of 500 mg will be administered intramuscularly (IM) into the buttocks slowly (1-2 minutes per injection) as two 5-mL injections, one in each buttock, on Days 1 and 15 of the run-in period.
  After the fulvestrant run-in, fulvestrant plus abemaciclib will be administered in 28-day cycles until disease progression or unacceptable toxicity. Fulvestrant (500 mg IM) will be administered on Day 1 of each 28-day cycle. Abemaciclib at a dose of 150 mg will be given p.o. BID on Days 1-28 of each cycle
  Interventions: Drug: Fulvestrant Run-In

INTERVENTIONS:
Drug: Fulvestrant Run-In — The study is evaluating if a drug holiday (post CDK inhibitors progression) will reset the cell cycle machinery to be responsive to Abemaciclib and Fulvestrant.
  Other Names: Abemaciclib; Fulvestrant

SUMMARY:
The study will investigate if CDK4/6 inhibitor holiday will reset the cell cycle process to respond to the combination of fulvestrant and abemaciclib, and this approach may represent an effective therapeutic strategy to manage such patients.

DETAILED DESCRIPTION:
Endocrine therapy, including aromatase inhibitor therapy, is the primary treatment for ER-positive metastatic disease. Despite the effectiveness of this treatment, not all patients respond to it and many patients who are initially responsive to the drug, eventually develop resistance to it. The management of patients with ER-positive, HER2-negative metastatic breast cancer who experience disease progression after standard treatment (CDK4/6 inhibitor plus an aromatase inhibitor) is a significant challenge and identification of new therapeutic strategies for this population of patients remains an unmet clinical need.

The aim of this research study is to determine if a month delay in the administration of the drug abemaciclib will be more effective than the drugs fulvestrant plus abemaciclib given together from the beginning for the treatment of ER-positive, HER2-negative metastatic breast cancer that has progressed on previous treatment. The study will investigate if a one month drug holiday from the CDK4/6 inhibitor drug, abemaciclib, will restore the body's sensitivity to the drug and make the subsequent treatment of abemaciclib plus fulvestrant more effective.

This is a single arm study where patients will receive fulvestrant for 1 month, followed by abemaciclib and fulvestrant every 28 days.

The treatment will be administered until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female >18 years of age on the day of informed consent signing.
2. Progression on a CDK4/6 inhibitor in combination with an AI immediately prior to the enrollment on this study
3. Histologically confirmed ER-positive, HER2-negative metastatic breast cancer. ER-positive is defined as ≥1% immunohistochemical (IHC) staining of any intensity. HER2 test result is negative if a single test (or both tests) performed show:

   * IHC 1+ or 0
   * In situ hybridization negative based on:

     * Single-probe average HER2 copy number <4.0 signals/cell
     * Dual-probe HER2/CEP17 ratio <2.0 with an average HER2 copy number <4.0 signals/cell.
4. Measurable disease according to the RECIST 1.1 or bone-only disease.
5. Postmenopausal status or receiving ovarian ablation with a gonadotropin-releasing hormone (GnRH) agonist. Postmenopausal status is defined by any one of the following criteria:

   * Prior bilateral oophorectomy
   * Age ≥55 years
   * Age <55 years and amenorrheic for at least 12 months (spontaneous cessation of menses for 12 consecutive months or more in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) and follicle-stimulating hormone and estradiol levels in the postmenopausal range without an alternative cause If the patient does not meet criteria for postmenopausal status but is receiving ovarian ablation therapy with a GnRH agonist, the patient is eligible for this trial, provided that the GnRH agonist is started at least 2 weeks prior to the first dose of trial treatment.
6. Eastern Cooperative Oncology Group performance status of 0 or 1.
7. Life expectancy ≥6 months.
8. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy). Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 21 days is required between end of radiotherapy and randomization.
9. Adequate organ function:

   * Absolute neutrophil count ≥1500/µL (without granulocyte colony stimulating factor support within 2 weeks of laboratory test used to determine eligibility)
   * Platelets ≥100,000/µL (without transfusion within 2 weeks of laboratory test used to determine eligibility)
   * Hemoglobin ≥9 g/dL (without blood transfusion)
   * White blood cell count >2,500/µL and <15,000/µL
   * Lymphocyte count ≥500/µL
   * Serum bilirubin ≤1.5x upper limit of normal (ULN; patients with known Gilbert's disease who have serum bilirubin level ≤3 x ULN may be enrolled)
   * Serum transaminases (aspartate transaminase [AST] or alanine transaminase [ALT]) activity ≤3.0 x ULN with normal alkaline phosphatase ([ALP]; patients with liver metastases ≤5 x ULN) OR AST and ALT ≤1.5 x ULN with ALP >2.5 x ULN
   * International normalized ratio and activated partial thromboplastin time ≤1.5 x ULN
   * Serum creatinine at or below the institutional normal value.
10. Able to swallow oral medication.
11. Patients who are made postmenopausal through use of GNRH agonists must be willing to use an adequate method of contraception for the course of the trial through 1 year after the last dose of trial treatment.
12. Patients who are made postmenopausal through use of GNRH agonists should have a negative serum pregnancy (β-human chorionic gonadotropin) within 7 days prior to trial treatment administration.
13. Willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of trial treatment administration.
2. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to trial treatment administration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to a previously administered agent. Note: If the patient received major surgery, she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting the trial treatment.
3. The patient has had major surgery within 14 days prior to starting the study.
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
6. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
7. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
8. Concurrent use of strong cytochrome P450 (CYP)3A inhibitors or inducers.
9. Hypersensitivity to fulvestrant, abemaciclib, or any of their excipients.
10. Manifestations of malabsorption due to prior gastrointestinal surgery, gastrointestinal surgery disease, or an unknown reason.
11. Has a bleeding disorder or currently taking anticoagulants.
12. Has active hepatitis B (detectable hepatitis B surface antigen) or active hepatitis C infection (detectable hepatitis C RNA).
13. Has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
14. Has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
15. Documented brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Patients with previously diagnosed brain metastases are eligible if they have completed treatment at least one month prior to trial treatment administration, are neurologically stable, and have recovered from effects of radiotherapy or surgery.

    * Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥2 weeks before trial treatment administration.
    * Treatment for brain metastases may have included whole brain radiotherapy, radiosurgery, or a combination as was deemed appropriate by the treating physician.
    * Patients who meet the above criteria and are clinically stable on anticonvulsant medication are eligible only if their anticonvulsant does not alter hepatic CYP activity in a way that might interfere with the metabolism of abemaciclib.
16. Have received any live vaccination within 28 days of trial treatment administration.
17. History within the last 12 months of any of the following conditions: syncope of cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest.
18. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) for fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant | TTF will be defined as time from start of therapy to discontinuation for any cause.
  Time to treatment failure (TTF) for fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant in patients with ER-positive, HER2-negative metastatic breast cancer that has progressed on a CDK4/6 inhibitor in combination with an AI, as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Estimation of the CBR of fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant | CBR will be defined as the percentage of patients with CR, PR, or stable disease (SD) according to the RECIST 1.1.
  Estimation of the CBR of fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant in patients with ER-positive, HER2-negative metastatic breast cancer that has progressed on a CDK4/6 inhibitor in combination with an AI, as assessed by the RECIST 1.1.
PFS rate between fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant. | PFS will be defined as the date of the first dose of trial treatment to the date of progression or death due to any cause, whichever occurs first, assessed up to 12 months after the last subject is added.
  PFS rate between fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant in patients with ER-positive, HER2-negative metastatic breast cancer that has progressed on a CDK4/6 inhibitor in combination with an AI.
Toxicity/safety between fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant. | Toxicity will be defined as any treatment-related death or any ≥ Grade 3 AE excluding alopecia and constitutional symptoms as assessed by the NCI CTCAE v4.03 through study completion, an average of 1 year.
  Toxicity/safety between fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant in patients with ER-positive, HER2-negative metastatic breast cancer that has progressed on a CDK4/6 inhibitor in combination with an AI, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Quality of life assessment after fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant. | Patient-reported quality of life after fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant, as assessed by the EORTC QLQ-C30 through study completion, an average of 1 year.
  Quality of life assessment after fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant in patients with ER-positive, HER2-negative metastatic breast cancer that has progressed on a CDK4/6 inhibitor in combination with an AI, as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30).
ORR of fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant. | ORR of fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant, as assessed by the RECIST 1.1 through study completion, an average of 1 year.
  ORR of fulvestrant plus abemaciclib with a 1-month run-in of fulvestrant in patients with ER-positive, HER2-negative metastatic breast cancer that has progressed on a CDK4/6 inhibitor in combination with an AI, as assessed by the RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Polly Niravath, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States